CLINICAL TRIAL: NCT03944967
Title: Postoperative Remote Monitoring of Vital Signs in Older Cardiac Surgery Patients
Acronym: AGEAWARE
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, PI, St. Antonius Hospital
Other Study IDs: NL68944.100.19
Record Dates: First submitted 2019-04-22; First posted 2019-05-10 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Hypoxemia; Respiratory Failure; Arrythmia
MeSH Terms: conditions — Hypoxia; Respiratory Insufficiency; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A significant number of elderly patients experience a complication after cardiac surgery. This study aims to determine if postoperative remote monitoring of vital signs can be used to identify medicatie risk factors for vital sign deterioration in older cardiac surgery patients.

* Single center pilot study.
* 100 older patients undergoing cardiac surgery.
* Continuous remote monitoring of vital signs after ICU discharge
* Main study endpoint is vital sign deterioration.

DETAILED DESCRIPTION:
Cardiac surgery in elderly patients aims to improve functional capacity and overall survival but may also precipitate major morbidity and mortality. Despite major improvements in the safety of anesthesia and surgery a significant number of elderly patients experience a complication after cardiac surgery.

To determine if postoperative remote monitoring of vital signs can be used to identify medication risk factors for vital sign deterioration in older cardiac surgery patients..

* Single center pilot study.
* 100 older patients undergoing cardiac surgery.
* Continuous remote monitoring of vital signs starts after ICU discharge
* PR, RR and SpO2 will be continuously monitored in all patients.
* Patients and healthcare personnel are blinded for monitoring results.
* Main study endpoint is vital sign deterioration.

The study population includes 100 patients ≥70 years undergoing elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years undergoing elective cardiac surgery.

Exclusion Criteria:

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes 100 patients ≥70 years undergoing elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | Three consecutive days after ICU discharge
  Duration of sPO2 <80%, <85%, <90% and <95% in minutes per hour
Respiratory deterioration | Three consecutive days after ICU discharge
  Duration of respiratory rate <10 min-1, >20 min-1, >25 min-1, >30 min-1 in minutes per hour
Arrythmia | Three consecutive days after ICU discharge
  Duration of pulse rate <50 min-1, >100 min-1, >110 min-1, >120 min-1 in minutes per hour

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided